CLINICAL TRIAL: NCT01358409
Title: Regression of Myocardial Steatosis by Nebivolol
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lidia Szczepaniak (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Lidia Szczepaniak, former Director of MR Spectroscopy laboratory, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTG_Neb01
Record Dates: First submitted 2011-05-20; First posted 2011-05-23 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Cardiac Steatosis and Lipotoxicity
Keywords: steatosis; MR spectroscopy; Nebivolol; cardiac MRI
MeSH Terms: conditions — Fatty Liver | interventions — Nebivolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nebivolol (Experimental): Nebivolol (Bystolic® by Forest/Mylan) is a third-generation beta-blocker; it selectively blocks β1-adrenergic receptors and increases peripheral vasodilation.
  Interventions: Drug: Nebivolol

INTERVENTIONS:
Drug: Nebivolol — Day 1 - Patients will start Nebivolol 5 mg PO daily; after one month, if the subject has tolerated 5 mg PO Nebivolol, the dose will be increased to 10 mg PO daily. If the patients is unable to tolerate 5 mg PO Nebivolol, he/she will be discontinued from the study. After six months, medication will be tapered to 5 mg PO daily for two weeks. Medication will then be tapered to 2.5 mg PO daily for two additional weeks.
  Other Names: Bystolic® by Forest/Mylan

SUMMARY:
Within large number of patients with obesity, it is crucial to determine who is at the greatest risk for development of chronic heart disease. The investigators previous studies suggest that an excessive accumulation of fat in heart cells precedes the development of obesity-related pathologies and may serve as a biomarker of heart disease in high-risk population. Until now, the evaluation of fat in the human heart was possible postmortem or by biopsy. The investigators novel magnetic resonance spectroscopy technique enables the quantification of intracellular lipid content non-invasively and repeatedly in humans in vivo. It could be used to better screen and treat obese patients at risk for the development of metabolic disease. The investigators hypothesize that in obese humans with elevated myocardial triglycerides, treatment with Nebivolol will reduce myocardial fat and will improve heart function.

DETAILED DESCRIPTION:
Background:

Epidemiological data have provided abundant evidence showing that obesity is a major risk factor for cardiovascular morbidity and mortality, although the exact mechanisms remain incompletely understood. Traditionally, obesity is thought to indirectly increase cardiovascular risk by means of its intermediary effects; obesity increases the risk of hypertension, dyslipidemia, and diabetes mellitus, thereby increasing one's overall risk for cardiovascular disease. In contrast to this traditional view, a growing body of research from our group and others advanced the novel hypothesis that ectopic myocardial fat deposition directly damages the heart. Lipid deposition and overload in the myocardium, termed "cardiac steatosis", is directly toxic to cardiac myocytes.

Deposition of lipid droplets in non-adipocytes (Steatosis): Normally, most of the triglycerides in the body are stored in adipose tissue with little to no lipid accumulation in non-adipocytes (e.g. parenchymal cells of the liver, pancreas, and muscle) due to a balance between fatty acid uptake and oxidation. When this mechanism is defective, fat accumulates in non-adipocytes. This abnormal retention of lipid within non-adipose tissues such as heart, liver, pancrease, and skeletal muscle is known as "steatosis" and reflects an impairment of the normal synthesis and elimination of triglyceride. This was first demonstrated in pancreatic β-cells of obese Zucker rats, a genetic model of obesity.

The intracellular accumulation of long chain free fatty acids (FFA) is hypothesized to engage an adverse signaling cascade in which conversion to Ceramide stimulates inducible nitric oxide synthase (iNOS), eventually leading to apoptosis. Progressive apoptosis of lipid-laden pancreatic β-cells over time eventually leads to insulin deficiency. A combination of β-cell failure and insulin resistance has produced diabetes in this animal model. More importantly, the pancreatic steatosis in pre-diabetic Zucker rats and the accompanying metabolic abnormalities were shown to be effectively reversed by the PPAR-Ƴ antagonist, Troglitazone.

The next logical step was to ask if similar mechanisms lead to deposition of lipid droplets within cardiomyocytes. Indeed, prediabetic obese Zucker rats deposit fat into cardiomyocytes; whereas, lean rats do not deposit fat in cardiomyocytes. Furthermore, the obese Zucker rats have progressive left ventricular systolic dysfunction, presumably due to excessive lipid deposition and toxicity, as dysfunction occurs before the onset of frank diabetes. In human studies, MR spectroscopy allows non-invasive evaluation of the number and size of lipid droplets in cardiomyocytes. Similar to the rodent studies, our group has demonstrated a strong linear relationship between triglyceride deposition in the myocardium and LV concentricity and function.

Nebivolol and its role in myocardial steatosis regression: Nebivolol (Bystolic® by Forest/Mylan)through its various modes of action has an exquisite ability to regress cardiac steatosis on many different levels. We propose a novel mechanism of Nebivolol action that results in reduction of myocardial steatosis.

Specific aims: This investigation will study whether: 1) cardiac steatosis plays a pivotal role in the early pathogenesis of obesity-related adverse cardiac remodeling in humans, 2) Nebivolol improves cardiac remodeling via its unique metabolic ability to reduce cardiac steatosis above and beyond its effect on hemodynamic cardiac remodeling due to blood pressure reduction.

Study Design and Hypotheses: Before and after six months of low dose (10 mg daily) Nebivolol treatment, localized proton MR spectroscopy (to measure triglyceride content in myocytes, as well as liver, pancreas and skeletal muscle) and cardiac MRI (for structural and functional measurements of the left ventricle) will be performed. Additionally, we will study abdominal subcutaneous fat levels over the six month period (MRI and Bioimpedance).

ELIGIBILITY:
Inclusion Criteria:

* Mexican American men and women
* Age 18 - 59
* Metabolic Syndrome*
* Myocardial TG > or = to 0.5% by localized MR spectroscopy

  *Metabolic syndrome in our study will follow the NCEP ATP III (National Cholesterol Education Program Adult Treatment Panel III) Guidelines which include > or = to 3 of the following:
* Fasting blood glucose > or = to 100 mg/dL
* Waist circumference: Men > 102 cm, Women > 88 cm
* Triglycerides > or = to 150 mg/dL
* BP > 130/85

Exclusion Criteria:

* Current use of a beta-blocker
* HR < 50 beats/min or BP < 130/85
* Contraindication to beta-blocker therapy such as asthma, reactive airway disease, heart block, or depression
* CHF (any NYHA class) by history, physical examination, or current use of CHF medication including beta-blockers, ACE inhibitors, angiotensin receptor blockers (ARBs), diuretics, calcium channel blockers, digitoxin, hydralazine, nitrates (including sublingual nitroglycerin), and inotropic agents
* LVEF < 50% by cardiac MRI
* Hepatic insufficiency or current use of another medication that is also metabolized by the CYP2D6 isozyme (paroxetine, fluoxetine, quinidine, propafenone).
* Any contraindication to MRI, e.g. metallic implants, metallic tattoos, claustrophobia, weight > 350 pounds (the MRI weight limit)
* Pregnancy at any time during the study
* A recent weight loss (>10% of body weight within the past year) or plans to undergo significant weight reduction (>10% of body weight) during the experimental protocol.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2011-04-01; Primary Completion 2013-02-11 (Actual); Study Completion 2013-02-11 (Actual)

PRIMARY OUTCOMES:
Myocardial triglyceride content | 6 months
  Regression of myocadial triglycerides using MR spectroscopy at two time points, one prior to receiving Nebivolol and six months after continuous low dose Nebivolol treatment.

SECONDARY OUTCOMES:
Cardiac function | 6 months
  Cardiac systolic and diastolic function will be assessed with cardiac MRI at two time points, one prior to receiving low dose Nebivolol treatment and once after six months of Nebivolol treatment.
Regression of concentric cardiac remodeling | 6 months
  Cardiac concentric remodeling will be assessed with cardiac MRI at two time points, one prior to receiving low dose Nebivolol treatment and once after six months of Nebivolol treatment.
Regression of steatosis in other non-adipocyte tissue | 6 months
  Regression of steatosis in other non-adipocyte tissue, including skeletal muscle, liver, and pancreas, will be assessed with MR spectroscopy at two time points, one prior to receiving low dose Nebivolol treatment and once after six months of Nebivolol treatment.
Regression of subcutaneous fat | 6 months
  Regression of subcutaneous fat will be assessed with cardiac MRI at two time points, one prior to receiving low dose Nebivolol treatment and once after six months of Nebivolol treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lidia S Szczepaniak, PhD, Principal Investigator — Cedars-Sinai Heart Institute
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States